CLINICAL TRIAL: NCT04824339
Title: Breast Cancer Endocrine Therapy FITness (BE-FIT) Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Kristin Campbell, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H20-03123
Record Dates: First submitted 2021-03-22; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Breast Neoplasms
Keywords: Exercise; Adjuvant endocrine therapy; Breast cancer survivor; Virtual Delivery; Reduce side effects
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): The intervention is an 8-week combined aerobic and resistance program, with virtual, group-based, supervised exercise sessions twice per week (60 min). The intervention also includes optional education on healthy eating.
  Interventions: Behavioral: Immediate Intervention Group
- Delayed Intervention Group (Experimental): Usual lifestyle control for 8 weeks and then invited to participate in the exercise intervention.
  Interventions: Behavioral: Delayed Intervention Group

INTERVENTIONS:
Behavioral: Immediate Intervention Group — This study is a partial cross over study. The intervention is 8 weeks in duration. Participants will be randomized to immediate exercise or delayed exercise, and the delayed exercise group will cross over to the intervention after 8 weeks.
  Arms: Immediate Intervention Group
Behavioral: Delayed Intervention Group — This study is a partial cross over study. The intervention is 8 weeks in duration. Participants will be randomized to immediate exercise or delayed exercise, and the delayed exercise group will cross over to the intervention after 8 weeks.
  Arms: Delayed Intervention Group

SUMMARY:
This project will assess the efficacy of an 8-week virtual exercise program on physical function offered to those with a breast cancer diagnosis currently receiving endocrine therapy. The intervention includes twice-weekly virtual group exercise classes. Participants also complete one to three independent home exercise sessions per week throughout the intervention. Testing will occur virtually at baseline, 8-weeks (at end of program) and follow-up evaluations will be performed at 16-weeks and 12- months after baseline testing. Questionnaires will be administered through REDCap. Exercise sessions and testing will be administered virtually via Zoom.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to test the effect of a virtually delivered supervised exercise program specific to breast cancer survivors on endocrine therapy versus delayed exercise in a partial cross over trial.

Justification: Endocrine therapy is commonly prescribed to breast cancer survivors for 5-10 years and often leads to side effects such as arthralgia, weight gain and bone density loss. Exercise has been shown to be an effective management strategy of these side effects and may improve quality of life and physical functioning. Many barriers exist surrounding the implementation of exercise programs for breast cancer survivors, despite the efficacious outcomes exercise programs have been shown to provide.

Due to COVID-19, virtual delivery options are needed to continue to provide exercise support to cancer patients. In September 2020, members of the investigator team successfully completed a pilot of the virtual intervention (n=30). In British Columbia, the investigators are well positioned to trial the implementation of an exercise program from a virtual setting, with programming specific to women receiving endocrine therapy. The knowledge gained from this study, if shown to be effective, will assist future program delivery and implementation across British Columbia for breast cancer survivors.

Aims and Objectives:

Primary Aim: To evaluate the efficacy of the exercise intervention group versus delayed exercise group to improve physical function, as measured by 30 second sit to stand test, from baseline to end of program (8-weeks).

Secondary Aim: To evaluate the preliminary efficacy of the intervention to improve endocrine therapy medication adherence (voils DOSE-non adherence measure) and endocrine symptom scores (FACT-ES) from baseline to end of program (8-weeks).

Tertiary Aim: To evaluate the preliminary efficacy of the intervention at improving exercise levels (modified Godin), health related quality of life (RAND), balance (tandem balance test) and self-reported anthropometric measures (weight, height, waist and hip circumference) from baseline to end of program (8-weeks).

Exploratory Aims: 1) To obtain additional data on efficacy outcomes (all outcomes listed above) with with-in group analysis of delayed exercise intervention group (0-8 weeks vs. 9-16 weeks) to further refine efficacy estimates to inform future implementation trials; and 2) to examine suitability of efficacy outcomes at 16-weeks (immediate intervention group only) and in both intervention arms, namely end of intervention 8- or 16-weeks, as appropriate to 12-months after baseline testing.

It is hypothesized that the intervention will improve physical function at 8 weeks. Additionally, it is hypothesized that the intervention will improve medication adherence, reduce self-reported endocrine symptoms, health-related quality of life, increase exercise levels, balance and anthropometrics at 8 weeks. The exploratory aims will provide information on maintenance effect in the short term (16 weeks) and longer term (12 months from enrollment).

Research Design: This study is a partial cross over study. The intervention is 8 weeks in duration. Participants will be randomized to immediate exercise or delayed exercise, and the delayed exercise group will cross over to the intervention after 8 weeks. This design was selected to optimize recruitment (all participants receive the intervention) while allowing appropriate comparison of intervention versus control, and to gain additional insights into efficacy of the intervention in order to better design future implementation studies. No washout period between crossover arms needed. Participants will undergo a virtual baseline assessment, 16 supervised virtual group-based exercise sessions delivered twice weekly, a final assessment at completion of the 8-week exercise program, as well as follow-up assessment at 16-weeks and 12-months after baseline testing. All sessions will take place virtually via a secure Zoom platform.

Statistical Analysis: Between group comparisons of those randomized to immediate intervention versus delayed intervention for changes in primary, secondary and tertiary outcomes from baseline to 8-weeks will be assessed using two-sample t-tests for normally distributed quantitative outcomes (primary, secondary, and tertiary). For highly skewed quantitative outcomes, the comparisons will be done using Mann-Whitney tests. For categorical outcomes, comparisons will use chi-square tests of independence (and Fisher Exact tests for binary outcomes).

For the delayed intervention group, within-group comparisons to assess changes from baseline (i.e., no intervention) to 16 weeks (i.e., after 8 weeks of delay plus 8 weeks of active intervention) will be done with paired t-tests for normally distributed outcomes, and Wilcoxon signed-rank tests for skewed quantitative outcomes.

A more formal repeated measures analysis of variance will be done to examine the change across multiple time points, which are baseline, 8 weeks, 16 weeks and 12-months. All tests will be two sided with a nominal level of significance of 5%.

An interim analysis will be undertaken once fifty percent of the planned sample size has been recruited and randomized. The aim of this analysis is to: 1) re-examine the target sample size using study data to compute effect size, and update if necessary; and 2) assess whether the trial should be stopped either due to tremendous efficacy or likely futility. This will be completed by the project statistician, and all other study team members will remain blinded, so that the randomization will not be jeopardized.

ELIGIBILITY:
Inclusion Criteria:

* Stage I - III breast cancer patients who are treated with curative intent
* Completed primary treatment, including surgery, radiation therapy and/or chemotherapy
* Currently receiving adjuvant endocrine therapy (Tamoxifen or an Aromatase Inhibitor) for at least 3 months (to allow for acclimatization) and within 3-years of of staring endocrine therapy.
* Can read and speak English
* Has access to a tablet, smartphone, laptop or computer with built-in video camera

Exclusion Criteria:

* Not currently receiving endocrine therapy or scheduled to stop within 6 months
* Diagnosed with stage IV breast cancer
* Not willing to attend a twice-weekly exercise program virtually for the duration of the study.
* Not willing to comply with safety measures of virtual programming (to be seen on camera and monitored via video by the instructor)

Ages: 19 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Function | Change from baseline to week 8 (end of intervention)
  Measured by 30 second sit to stand test

SECONDARY OUTCOMES:
Medication adherence to endocrine therapy | Change from baseline at week 8 (end of intervention), 16 weeks and 12-months
  Measured by Voils DOSE-non adherence measure; where higher scores indicate greater levels of nonadherence.
Health-related quality of life | Change from baseline at week 8 (end of intervention), 16 weeks and 12-months
  Measured by RAND 36-Item Short Form Health Survey
Usual physical activity levels | Change from baseline at week 8 (end of intervention), 16 weeks and 12-months
  Modified Godin Leisure Time Physical Activity questionnaire
Weight in kilograms | Change from baseline at week 8 (end of intervention), 16 weeks and 12-months
  Measured using a scale in kilograms
Height in metres | Change from baseline at week 8 (end of intervention), 16 weeks and 12-months
  Measured using stadiometer in metres
Body mass index | Change from baseline at week 8 (end of intervention), 16 weeks and 12-months
  Aggregated measure of height and weight, reported in kg/m^2
Waist circumference | Change from baseline at week 8 (end of intervention), 16 weeks and 12-months
  Measures circumference in centimeters
Hip circumference | Change from baseline at week 8 (end of intervention), 16 weeks and 12-months
  Measures circumference in centimeters
Standing balance | Change from baseline at week 8 (end of intervention), 16 weeks and 12-months
  Tandem balance test measured in seconds
Physical Function | Change from baseline at week 8 (end of intervention), 16 weeks and 12-months
  Measured by 30 second sit to stand test

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Campbell, PhD, Principal Investigator — Department of Physical Therapy
Locations (1):
- Clinical Exercise Physiology Lab, Vancouver, British Columbia, Canada